CLINICAL TRIAL: NCT00653198
Title: Hospital-based, Case-control Study to Assess the Vaccine Effectiveness of Rotarix™ Against Rotavirus Severe Gastroenteritis (RV SGE) Among Hospitalised Children Born After 1 March 2006 and at Least 12 Weeks of Age, in Panama
Brief Title: Effectiveness of Rotarix™ Against Rotavirus Severe Gastroenteritis (RV SGE) in Infants in Panama
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 104676
Record Dates: First submitted 2008-03-19; First posted 2008-04-04 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Infections, Rotavirus
Keywords: Rotavirus severe gastroenteritis (RV SGE)
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples

GROUPS / COHORTS (2):
- A: Cases
  Interventions: Other: No intervention
- B: Controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This study aims to estimate the effectiveness of Rotarix™ vaccine which is used nationwide as a part of the expanded program on immunization (EPI), in preventing RV SGE among hospitalised children born after 1 March 2006, which corresponds to the date of introduction of Rotarix™ in the national immunization program.

ELIGIBILITY:
Inclusion Criteria for enrolled subjects and cases :

* A male or female child born after 1 March 2006 (which corresponds to the date of introduction of Rotarix™ in the EPI) and at least 12 weeks of age.
* Subject admitted to the study hospital for SGE (refer to the glossary) during the study period.
* Onset of SGE <= 14 days prior to admission.
* Laboratory confirmed (i.e. by ELISA at the hospital laboratory) RV positive stool sample at hospital admission or during the first 48 hours of hospitalisation. Note: This criterion is applicable only for cases.
* Written informed consent obtained from the parent or guardian of the subject.

Inclusion criteria for controls:

* Admitted for non-GE causes at the same hospital as the case. Note: This criterion is applicable to hospital controls only.
* Living in the same neighbourhood as the case for at least three consecutive months. Note: This criterion is applicable to neighbourhood controls only.
* At least 12 weeks of age and being born within ± 2 weeks from the date of birth of the case. If the list of children born within ± 2 weeks is exhausted, then the range would be extended to ± 4 weeks.
* Written informed consent obtained from the parent or guardian of the child.

Exclusion Criteria for enrolled subjects and cases:

* Subject has previously participated as case or control in this study.
* Hospitalisation is unrelated to GE.
* Onset of SGE > 48 hours after admission to the hospital (nosocomial infections).

Exclusion criteria for controls:

* For hospital controls: Child who has symptoms of GE during current hospitalisation or on the day of interview of his/her parent or guardian.

OR

* For neighbourhood controls: Child who has symptoms of GE on the day of interview of his/her parent or guardian.
* Exclude children with the following vaccine preventable diseases: measles, mumps, rubella, diphtheria, pertussis, tetanus, tuberculosis, invasive Haemophilus Influenzae Type B (Hib) infections (meningitis, bacteraemia, septic arthritis, cellulitis, and epiglottitis) and hepatitis B.
* Child has participated in the past as a case or control in this study.
* Child living in the same house as the case. Note: This criterion is applicable to neighbourhood controls only

Min Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases will include those children born after 1 March 2006, at least 12 weeks of age and hospitalised for RV SGE in the study hospital, during the designated study period. For each case, three hospital controls and three neighbourhood controls will be included in the study, after matching by date of birth. Hospital controls will be children hospitalised for non-GE causes in the study hospital during the same time period as the case. Neighbourhood controls will be children without any symptoms of GE or SGE, and residing in the same area as the case at least for three consecutive months.
Sampling Method: Probability Sample
Enrollment: 885 (Actual)
Dates: Start 2008-03-19 (Actual); Primary Completion 2011-03-18 (Actual); Study Completion 2011-03-18 (Actual)

PRIMARY OUTCOMES:
Occurrence of RV GE among children born after 1 March 2006, at least 12 weeks of age and admitted to the study hospital for SGE.

SECONDARY OUTCOMES:
Occurrence of acute GE among children born after 1 March 2006, at least 12 weeks of age and admitted to the study hospital for SGE.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Panama City, Panama